CLINICAL TRIAL: NCT06763393
Title: Correlation Between Adnexal Masses and Endometrial Thickness Measured With Ultrasound in Adults Women
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/036
Record Dates: First submitted 2024-12-18; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Endometrial Disorder
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Ultrasound — To determine the correlation between adnexal masses and endometrial thickness measured with ultrasound in adults women.

SUMMARY:
This study explores the correlation between adnexal masses and endometrial thickness in adult women, using ultrasound as the primary diagnostic tool.

DETAILED DESCRIPTION:
Adnexal masses, including ovarian cysts and other abnormalities, are common gynecological findings, while endometrial thickness is a crucial indicator for assessing conditions like endometrial hyperplasia or malignancy.

By analyzing ultrasound data, this research aims to determine whether the presence, size, or characteristics of adnexal masses have a significant relationship with variations in endometrial thickness.

ELIGIBILITY:
Inclusion Criteria:

* Adult women typically defined as those aged 18 and older.
* Women with diagnosed adnexal masses, which could be cysts, tumors, or other growths in the adnexa (ovaries and fallopian tubes).

Exclusion Criteria:

* Pregnant women might have different hormonal and physiological changes that can affect endometrial thickness and adnexal masses.
* Recent gynecological history.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adnexal Masses and Endometrial Thickness
Study Population: to check the Correlation Between Adnexal Masses and Endometrial Thickness Measured With Ultrasound
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
ultrasound for Endometrial Thickness | 12 Months
  Endometrial thickness is well assessed on MRI. Measurement should be taken at a mid-sagittal slice, similar to the ultrasound assessment plane
ultrasound radiopaedia for Adnexal Masses | 12 months
  Ultrasound (US) is an imaging technology that uses high-frequency sound waves to characterize tissue. It is a useful and flexible modality in medical imaging and often provides an additional or unique characterization of tissues

CONTACTS AND LOCATIONS:
Locations (1):
- Sadiqabad, Sadiqābād, Punjab Province, Pakistan